CLINICAL TRIAL: NCT00561626
Title: Effects of a High-fat and a Low-fat Diet on Early Biomarkers of Metabolic Stress in Blood and Gene Expression in the Small Intestine of Healthy Subjects
Brief Title: Effects of High-fat and Low-fat Diet on the Gut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Ronald P. Mensink, Prof. Dr. Ir., Maastricht University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 07-3-088
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2008-12

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Dietary Supplement: high fat diet followed by low fat diet
- B (Experimental)
  Interventions: Dietary Supplement: low fat diet followed by high fat diet

INTERVENTIONS:
Dietary Supplement: high fat diet followed by low fat diet — High fat diet : 40 Energy (En)% fat, 45 En% carbohydrates, 15 En% proteins, 250 mg cholesterol,4 weeks, daily Low fat diet : 20 Energy (En)% fat, 65 En% carbohydrates, 15 En% proteins, 250 mg cholesterol,4 weeks, daily
  Arms: A
Dietary Supplement: low fat diet followed by high fat diet — Low fat diet : 20 Energy (En)% fat, 65 En% carbohydrates, 15 En% proteins, 250 mg cholesterol,4 weeks, daily High fat diet : 40 Energy (En)% fat, 45 En% carbohydrates, 15 En% proteins, 250 mg cholesterol,4 weeks, daily
  Arms: B

SUMMARY:
Rationale: The prevalence of the metabolic syndrome is strongly increasing in developed countries. The role of the small intestine seems important in the development of the metabolic syndrome. Although it is known that a high-fat Western-style of diet has deleterious effects on (post-prandial) lipidemia and glucose homeostases, effects of such a diet on the small intestine is not known. To elucidate the role of the small intestine on the early development of the metabolic syndrome, the effects of a high-fat (HF) and a low-fat (LF) diet will be examined on gene expression in the small intestine and early biomarkers in blood of healthy subjects.

Objective: The objective of this study is to compare in healthy subjects the effects of a HF diet (40 En% fat) with those of a LF diet (20 En% fat) on early biomarkers and parameters of metabolic stress in blood and on expression of genes in the small intestine.

Additional research objectives are:

* To compare the diet-induced changes in transcriptome profile of the small intestine with more easily accessible peripheral blood mononuclear cells (PBMC)
* To establish effects of HF and LF diet on basal gut permeability and after a chenodeoxycholic acid (CDCA) load (second hit).

Study design: Randomised crossover design. The duration of the experimental periods (HF and LF diet) will be 28 days, separated by a wash out period of at least 3 weeks. At day 21 of each intervention period a postprandial test will be performed and duodenum biopsies will be taken. At day 25 and 28 of each intervention period, respectively, basal gut permeability and gut permeability after a CDCA load will be determined with a sugar recovery test.

Study population: Ten healthy men in the age of 18-60 years, without a history of any gastrointestinal disorders or complaints.

Intervention: Subjects will consume in random order:

* a HF diet (40 En% fat, 45 En% carbohydrates and 15 En% proteins)
* a LF diet (20 En% fat, 65 En% carbohydrates and 15 En% proteins)

Primary study parameters/endpoints: Potential early biomarkers of the metabolic syndrome in blood and gene expression profiles in the small intestine.

Secondary study parameters/endpoints: Parameters of the metabolic syndrome in blood, gene expression profiles in PBMC and gut permeability.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* body mass index (BMI) between 18 and 30 kg/m2

Exclusion Criteria:

* BMI ≤ 18 and ≥ 25 kg/m2
* Smoking
* Serum Total cholesterol > 8.0 mmol/L
* Fasting glucose > 7.0 mmol/L
* Use of any medication
* Active cardiovascular diseases like congestive heart failure or recent (<6 months) event (acute myocardial infarction, CVA)
* Gastrointestinal diseases (like celiac disease, inflammatory bowel disease, irritable bowel disease and food allergies) or a history of any gastrointestinal disorders or complaints
* Pre-existing gallbladder disease
* Diabetes mellitus
* Familial hypercholesterolemia
* Severe medical conditions that might interfere with the study such as epilepsy, asthma, COPD and rheumatoid arthritis.
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Impairment of renal function, as evidenced by increased serum creatinine >150 mmol/L
* Hepatic diseases as manifested by ALT, AST, GGT, total bilirubin or ALP > 2 times the upper limit of normal
* CRP values > 8.0 mg/mL
* Abuse of drugs and/or alcohol
* Participation in another biomedical study within 1 month prior to the start of this study
* Having donated blood (as blood donor) within 1 month prior to start of this study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
potential early biomarkers in plasma | 3 weeks

SECONDARY OUTCOMES:
gene expression in the small intestine and in peripheral blood mononuclear cells (PBMC) | 3 weken
gut permeability | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P. Mensink, Prof. Dr. Ir., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Department of Human Biology, Maastricht, Netherlands